CLINICAL TRIAL: NCT02923687
Title: Premedication Efficacy of Ketorolac Infiltration on Post Endodontic Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azad University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Nahid Mohammadzadeh Akhlaghi, Associate Professor, Azad University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: AZadUMS-P/190/D
Record Dates: First submitted 2016-09-29; First posted 2016-10-04 (Estimated); Last update posted 2019-01-15 (Actual); Status verified 2019-01

CONDITIONS: Irreversible Pulpitis
Keywords: Ketorolac; Root canal treatment; Pain; Premedication
MeSH Terms: conditions — Pain | interventions — Ketorolac Tromethamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buccal infiltration of Ketorolac (Active Comparator): All patients will receive standard inferior alveolar nerve block of 2% lidocaine with 1:800000 epinephrine and supplemental buccal infiltration of 0.9 mL 2% lidocaine with 1:800000 epinephrine. After five minutes, case group will receive a supplemental buccal infiltration of 30 mg/mL of Ketorolac tromethamine (Alborz-Darou Co. Qazvin, Iran).
  Interventions: Drug: Ketorolac Tromethamine
- Buccal infiltration of Normal saline (Placebo Comparator): All patients will receive standard inferior alveolar nerve block of 2% lidocaine with 1:800000 epinephrine and supplemental buccal infiltration of 0.9 mL 2% lidocaine with 1:800000 epinephrine. After five minutes, the control group will receive normal saline as placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ketorolac Tromethamine — All patients will receive standard inferior alveolar nerve block of 2% lidocaine with 1:800000 epinephrine and supplemental buccal infiltration of 0.9 mL 2% lidocaine with 1:800000 epinephrine. After five minutes, the experimental group will receive supplemental buccal infiltration of 30 mg/mL of Ketorolac Tromethamine.
  Other Names: Tradol Alborz-Darou Co. Qazvin, Iran
  Arms: Buccal infiltration of Ketorolac
Drug: Placebo — All patients will receive standard inferior alveolar nerve block of 2% lidocaine with 1:800000 epinephrine and supplemental buccal infiltration of 0.9 mL 2% lidocaine with 1:800000 epinephrine. After five minutes, control group will receive buccal infiltration of normal saline.
  Other Names: Normal saline
  Arms: Buccal infiltration of Normal saline

SUMMARY:
Objective: The aim of this study is to evaluate premedication with ketorolac infiltration on post endodontic pain in patients with symptomatic irreversible pulpitis.

Design: Randomized double blind clinical trial

Setting and conduct: Sixty adult volunteers with including criteria will be divided into two groups (n=30) based on random table. All patients will receive standard inferior alveolar nerve block of 2% lidocaine with 1:800000 epinephrine and supplemental buccal infiltration of 0.9 mL 2% lidocaine with 1:800000 epinephrine. After five minutes one group will receive supplemental buccal infiltration of 30 mg/mL of Ketorolac Tromethamine and the control group will receive buccal infiltration of normal saline. Endodontic access preparation will initiate after 15 minutes of initial IANB with two negative responses to the electric pulp test. The pain level will be recorded immediately and at the 2,4,6 and 24 hours following the treatment using Heft- Parker Visual Analog Scale (HP- VAS). Data will be evaluated using Repeated measured test (if possible) and otherwise non-parametric tests such as rival Friedman and X2 test. Participants including major eligibility criteria: all patients age ranged 18-65 with symptomatic irreversible pulpitis (HP VAS ≥54) and without pain on percussion on a mandibular molar tooth who need root canal treatment and are without systemic diseases; nonsmoking; non pregnant, non breast feeding without any medicine consumption or analgesic and sedation

Intervention: Ketorolac infiltration

Main outcome measures: Pain level at immediately after the treatment, 2, 4, 6 and 24 hours following the root canal treatment using HP VAS.

DETAILED DESCRIPTION:
Objective: The aim of this study is to evaluate premedication with ketorolac infiltration on post endodontic pain in patients with symptomatic irreversible pulpitis.

Design: Randomized double blind clinical trial

Setting and conduct: Sixty adult volunteers with including criteria will be divided into two groups (n=30) based on random table. All patients will receive standard inferior alveolar nerve block of 2% lidocaine with 1:800000 epinephrine and supplemental buccal infiltration of 0.9 mL 2% lidocaine with 1:800000 epinephrine. After five minutes one group will receive supplemental buccal infiltration of 30 mg/mL of Ketorolac Tromethamine and the control group will receive buccal infiltration of normal saline. Endodontic access preparation will initiate after 15 minutes of initial IANB with two negative responses to the electric pulp test. Endodontic treatment of all the patients will be performed in a single visit, using crown down method and with rotary instrumentation till master apical file size# 30.06. The pain level will be recorded immediately and at the 2,4,6 and 24 hours following the treatment using Heft- Parker Visual Analog Scale (HP- VAS). Data will be evaluated using Repeated measured test (if possible) and otherwise non-parametric tests such as rival Friedman and X2 test. Participants including major eligibility criteria: all patients age ranged 18-65 with symptomatic irreversible pulpitis (HP VAS ≥54) and without pain on percussion on a mandibular molar tooth who need root canal treatment and are without systemic diseases; nonsmoking; non pregnant, non breast feeding without any medicine consumption or analgesic and sedation

Intervention: Ketorolac infiltration

Main outcome measures: The pain level immediately and at the 2, 4, 6 and 24 hours following the treatment using HP- VAS

ELIGIBILITY:
Inclusion Criteria:

* patients with age ranged 18-65;
* without systemic diseases;
* without any medicine consumption;
* non smoking;
* non pregnant;
* non breast feeding;
* with symptomatic irreversible pulpitis (Visual Analog Scale ≥ 54) in one mandibular molar without apical periodontitis that needs root canal treatment.

Exclusion Criteria:

* The patients less than 18 and more than 65 years old;
* systemic diseases;
* any medicine consumption;
* smoking;
* pregnant;
* breast feeding;
* apical periodontitis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Premedication effect of Ketorolac buccal infiltration on post Endodontic pain | 24 hours
  The pain level after the root canal therapy will be recorded using HP-VAS up to 24 hours in each of the case and control groups and will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Nahid Mohammadzadeh Akhlaghi, DDS,MDS, Study Chair — Associate Professor
Locations (1):
- Dental Branch, AZad UMS, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Yes